CLINICAL TRIAL: NCT01491334
Title: A Clinical Validation Study With Transvaginal Tactile Imaging
Brief Title: Validation of Transvaginal Tactile Imaging
Acronym: VTI-03
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: VTI-03; 1R43AG034714 (NIH)
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: POP; Pelvic Floor; Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asymptomatic: Asymptomatic women presenting at various ages without prolapse condition.
- Symptomatic: Symptomatic women presenting with prolapse conditions with no prior surgeries and women presenting with surgery scheduled with or without prior surgery.

SUMMARY:
The purpose of this study is to validate safety and effectiveness in assessment of the female pelvic floor tissue, and, assess the ability of Vaginal Tactile Imager (VTI) to detect early prolapse conditions and characterize the outcome of reconstructive surgery.

DETAILED DESCRIPTION:
1. The device will detect significant differences in tissue elasticity and anatomy for women with normal pelvic floor versus women with prolapse stage 1.
2. The device will detect significant differences in tissue elasticity and anatomy for patients before and after reconstructive surgery.
3. The device will detect significant differences in tissue elasticity and anatomy among 3 groups of patients with prolapse stages 1, 2 and 3.
4. The device will detect significant differences in tissue elasticity among 3 control groups with normal pelvic floor conditions (nulliparous women at age 21-30, parous women at age 31-40, and postmenopausal women).

ELIGIBILITY:
Inclusion Criteria:

* Subject is female of 21 years or older AND HAS AT LEAST ONE OF THE FOLLOWING
* No evidence of pelvic organ prolapse and no prior pelvic surgery
* Stage 1 or greater pelvic organ prolapse affecting one or more vaginal compartments and no prior pelvic surgery
* Stage 2 or greater pelvic organ prolapse affecting one or more vaginal compartments and reconstructive surgery is scheduled

Exclusion Criteria:

* Active skin infection or ulceration within the vagina
* Presence of a vaginal septum;
* Active cancer of the colon, rectum wall, cervix, vaginal, uterus or bladder;
* Ongoing radiation therapy for pelvic cancer;
* Impacted stool
* Recent (less than three months) pelvic surgery;
* Significant pre-existing pelvic pain including levator ani syndrome, severe vaginismus or vulvodynia;
* Severe hemorrhoids
* Surgically absent rectum or bladder
* Significant circulatory or cardiac conditions that could cause excessive risk from the examination as determined by attending physician

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient pool will comprise of 200 female patients.
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2011-12; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Effectiveness in assessment of the pelvic floor tissue conditions. | Two years.
Ability in early detection of prolapse conditions. | One Year
Ability in characterization of the outcome of pelvic floor reconstructive surgery. | Two years.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Egorov, Ph.D., Principal Investigator — Artann Laboratories, Inc.
Locations (2):
- United States (2):
  - Princeton Urogynecology, Princeton, New Jersey
  - Institute of Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania

REFERENCES:
- [Result] Sarvazyan A, Egorov V. Mechanical Imaging - a Technology for 3-D Visualization and Characterization of Soft Tissue Abnormalities. A Review. Curr Med Imaging Rev. 2012 Feb 1;8(1):64-73. doi: 10.2174/157340512799220571. PMID 24058326
- [Result] van Raalte H, Egorov V, Lucente V, Murphy M, Saiz C. 3D tactile imaging in early prolapse detection. International Continence Society 43rd Annual Meeting. Barcelona, Spain, 26-30 August, 2013.
- [Result] Egorov V, van Raalte H, Lucente V. Tactile imaging and tissue elasticity as a marker of pelvic floor conditions. International Urogynecological Association: 38th Annual Meeting, Dublin, Ireland, May 28-June 1, 2013.
- [Result] van Raalte H, Lucente V, Egorov V. Measuring outcome in urogynecological surgery by 3-D tactile imaging: First clinical experience. International Urogynecological Association: 38th Annual Meeting, Dublin, Ireland, May 28-June 1, 2013.
- [Result] van Raalte H, Egorov V, Lucente V. Tissue elasticity as a marker of pelvic floor conditions: Clinical results. Proceedings of the 11th International Tissue Elasticity Conference, Deauville, France, October 2-5, 2012: 46.